CLINICAL TRIAL: NCT04512924
Title: Food Allergy Symptom Self-management With Technology (FASST) for Caregivers: An mHealth Intervention to Address Psychosocial Outcomes in Caregivers of Children With Newly Diagnosed Food Allergy
Brief Title: The Psychosocial Outcomes in Caregivers of Children With Food Allergy
Acronym: FASST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00100789
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Food Allergy in Children; Caregiver Burnout; Psychosocial Problem; Family Research
MeSH Terms: conditions — Caregiver Burden | interventions — Standard of Care; Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Behavioral: Enhanced mobile app with standard of care and education
- Group 2 (Experimental)
  Interventions: Behavioral: Enhanced mobile app with standard of care, education and support resources

INTERVENTIONS:
Behavioral: Enhanced mobile app with standard of care and education — Group 1 will download an enhanced mobile app that will include education and support resources related to food allergy and its management.
  Arms: Group 1
Behavioral: Enhanced mobile app with standard of care, education and support resources — Group 2 will download an enhanced mobile app that will include education and support resources related to food allergy and its management, a symptom monitoring and tracking system that allows mobile app users to log symptoms they may experience as caregivers of children newly diagnosed with food allergy, e.g. fatigue and anxiety, and symptom based interventions (recommendations) that may improve a caregiver's ability to self-manage experienced symptoms.
  Arms: Group 2

SUMMARY:
The purpose of this study is to evaluate use of a mobile application (also commonly referred to as an app) designed to support caregivers of children with newly diagnosed food allergy. This study has 2 phases. In Phase 1, the researchers obtained feedback regarding use of mobile apps from caregivers who have been managing their child's food allergy for one year or more. The researchers then used this feedback to build a mobile app for caregivers of children with newly diagnosed food allergy. In Phase 2, the researchers will evaluate the mobile app during a 4-week evaluation period with a group of caregivers of children newly diagnosed with food allergy. The data obtained from this study will hopefully benefit caregivers of children with newly diagnosed food allergy.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of child less than or equal to 18 years of age who are newly diagnosed (less than or equal to 90 days from diagnosis) with food allergy(ies).

Exclusion Criteria:

* Caregiver with cognitive impairment/deficit and/or observed lack of understanding during the informed consent process

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Broome SB, Williams KW, Hendrix KH. App providing psychosocial and educational supports benefits caregivers of children with newly diagnosed food allergies. J Food Allergy. 2022 Dec 1;4(3):163-171. doi: 10.2500/jfa.2022.4.220035. eCollection 2022 Dec. PMID 39036772
- [Derived] Broome B, Madisetti M, Prentice M, Williams KW, Kelechi T. Food Allergy Symptom Self-Management With Technology (FASST) mHealth Intervention to Address Psychosocial Outcomes in Caregivers of Children With Newly Diagnosed Food Allergy: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2021 Mar 3;10(3):e25805. doi: 10.2196/25805. PMID 33656448

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 20 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34 [27 to 43] | 32.3 [19 to 42] | 33.1 [19 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 20 | 29
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 10 | 17 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 7 | 14 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Fatigue as Assessed by Patient-Reported Outcomes Measurement Information System Fatigue Short Form: PROMIS Short Form 6a
Description: The PROMISED Interference (Short Form 6a) instrument measures the self-reported consequences of fatigue across aspects of life including social, cognitive, emotional, physical and recreational activities; this instrument refers to the past seven days. This validated scale has five response options, with scores ranging from one to five. Scores are converted to t-scores, and higher t-scores indicate greater pain interference. Higher scores represent greater degrees of fatigue. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe fatigue. Fatigue T-scores measured by PROMIS Fatigue Short Form 6a. This 6-item instrument assesses a patient's a patient's level of fatigue over a 7-day recall period. Respondents report fatigue on a 5-point scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 33.4 to 76.8. Lower T-scores represent better outcomes.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
score on a scale | 50.6 [43.3 to 57.8] | 53 [48.5 to 57.4]

2. Primary Outcome: Fatigue as Assessed by Patient-Reported Outcomes Measurement Information System Fatigue Short Form. PROMIS Short Form 6a
Description: The Patient-Reported Outcomes Measurement Information System Fatigue item banks assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe fatigue. Fatigue T-scores measured by PROMIS Fatigue Short Form 6a. This 6-item instrument assesses a patient's a patient's level of fatigue over a 7-day recall period. Respondents report fatigue on a 5-point scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 33.4 to 76.8. Lower T-scores represent better outcomes.
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
score on a scale | 52.2 [48.1 to 56.3] | 49.5 [46.1 to 53]

3. Primary Outcome: Sleep Disturbance as Assessed by Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form. PROMIS Sleep Disturbance Short Form 6a
Description: Change in mean sleep disturbance score measured with PROMIS Sleep Disturbance short form 6a, 6 individual items allow for different responses which are scored separately to provide specific information about self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. The lowest possible raw score is 6; the highest possible raw score is 30. Raw summed scores are converted to T-score values that are standardized such that 50 represents the average (mean) for the US general population, and a standard deviation of 10 points. A higher T-score represents more of the concept being measured, meaning the higher above 50 the worse or the greater the individual's sleep is disturbed compared to individuals with chronic conditions. Scores <55 within normal limits, 55-60 mild, 61-70 moderate, >70 severe sleep disturbance.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
score on a scale | 59.9 [58 to 61.8] | 58.8 [57 to 60.6]

4. Primary Outcome: Sleep Disturbance as Assessed by Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form. PROMIS Sleep Disturbance Short Form 76a
Description: The Patient-Reported Outcomes Measurement Information System Sleep Disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. A low score indicates low sleep disturbance; high score indicates high sleep disturbance. Scores less than 55 are "within normal limits," 55-60 are "mild," 60-70 are "moderate," and greater than 70 are "severe." Raw scores on the survey are converted to T scores, which are standardized scores based on the average in the population; a score of 50 would indicate meeting the T score for the average quality of sleep in the reference general population, with a standard deviation of 10. Higher T scores reflect greater sleep disturbance, and thus worse outcomes. The means reported are the mean T scores at the indicated timepoint.
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
score on a scale | 59.3 [57.1 to 61.5] | 59.7 [58 to 61.4]

5. Primary Outcome: Depression as Assessed by Patient-Reported Outcomes Measurement Information System Depression Short Form. PROMIS Depression Short Form 6a
Description: The Patient-Reported Outcomes Measurement Information System Depression item banks assess self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Higher scores indicate negative mood; lower scores indicate more positive mode. Six items are rated on a 5 point scale that assess caregiver depression; 1=Never to 5=Always. To find the total raw score, sum the values of the response to each question. Higher scores indicate greater severity in depression. Scores less than 55 are "within normal limits," 55-60 are "mild," 60-70 are "moderate," and greater than 70 are "severe." T-score range 38 to 81; 50 indicates the population mean with a standard deviation of 10; minimally important difference greater than or equal to 3 points; higher scores indicate worse outcome.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
T-score | 43.6 [37.6 to 49.6] | 45.9 [42.2 to 49.6]

6. Primary Outcome: Depression as Assessed by Patient-Reported Outcomes Measurement Information System Depression Short Form. PROMIS Depression Short Form 6a
Description: as for outcome 5
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
T-score | 44.1 [39.5 to 48.7] | 45.6 [41.2 to 50]

7. Primary Outcome: Anxiety as Assessed by Patient-Reported Outcomes Measurement Information System Anxiety Short Form. PROMIS Anxiety Short Form 6a
Description: The Patient-Reported Outcomes Measurement Information System Anxiety item banks assess self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). The anxiety measure is universal rather than disease-specific. Higher scores indicate higher levels of anxiety; lower scores indicate lower levels of anxiety. Six items are rated on a 5 point scale that assess caregiver anxiety; 1=Never to 5=Always. To find the total raw score, sum the values of the response to each question. Higher scores indicate a greater severity in anxiety. Scores less than 55 are "within normal limits", 55-60 are "mild", 60-70 are "moderate", and greater than 70 are "severe". The raw score is converted to a T-score ranging from 31.7 to 76.1. 50 indicates the population mean with a standard deviation of 10. Higher T-scores indicate greater anxiety disturbance.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
T-score | 51.2 [42.8 to 59.5] | 55.1 [50 to 60.3]

8. Primary Outcome: Anxiety as Assessed by Patient-Reported Outcomes Measurement Information System Anxiety Short Form. PROMIS Anxiety Short Form 6a
Description: The Patient-Reported Outcomes Measurement Information System Anxiety item assess self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness) . The anxiety measure is universal rather than disease-specific. Higher scores indicate higher levels of anxiety; lower scores indicate lower levels of anxiety. Six items are rated on a 5 point scale that assess caregiver anxiety; 1=Never to 5=Always. To find the total raw score, sum the values of the response to each question. Higher scores indicate a greater severity in anxiety. Scores less than 55 are "within normal limits", 55-60 are "mild", 60-70 are "moderate", and greater than 70 are "severe". The raw score is converted to a T-score ranging from 31.7 to 76.1, 50 indicates the population mean with a standard deviation of 10 Higher T-scores indicate greater anxiety disturbance.
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
T-score | 51.2 [44.7 to 57.6] | 52.3 [47.8 to 56.8]

9. Primary Outcome: Caregiver Self-efficacy Related to Managing Food Allergy in Child as Assessed by the Food Allergy Self-Efficacy Scale for Parents:(FASE-P): Treat my Child if They Had an Allergic Reaction
Description: Food Allergy Self Efficacy Scale for Parents (FASE-P) The FASE-P measures parental confidence in their ability to manage their child's FA. Subdomains include managing social activities, precaution and prevention, allergic treatment, food allergen identification, and seeking information about FA. Each item is rated from 0-100 and a mean score is calculated. Higher scores indicate greater FA-related self-efficacy. The FASE-P offers excellent reliability over time in a general FA population.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
score on a scale | 78.7 [61.8 to 95.6] | 87.2 [78.2 to 96.2]

10. Primary Outcome: Caregiver Self-efficacy Related to Managing Food Allergy in Child as Assessed by the Food Allergy Self-Efficacy Scale for Parents (FASE-P):Treat my Child if They Had an Allergic Reaction
Description: as for outcome 9
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
score on a scale | 86.5 [74.9 to 98.1] | 92.6 [87.5 to 97.8]

11. Primary Outcome: Change in Caregiver Quality of Life-parental Burden as Assessed by the Food Allergy Quality of Life-Parental Burden (FAQoL-PB): How Limited Would Your Ability to Participate in Social Activities That Involve Food be Because of Your Child's Food Allergy?
Description: The FAQL-PB is a 17-item questionnaire designed to capture caregiver HRQoL in children ages 0-12 years with FA. Items are rated on a 7-point Likert scale (0=not limited/troubled to 6=extremely limited/troubled); a mean score is calculated with higher scores indicating poorer HRQoL.
Time Frame: Baseline and 30 days
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
score on a scale | 2.9 [1.8 to 4.0] | 2.8 [2.0 to 3.6]

12. Primary Outcome: Change in Caregiver Quality of Life-parental Burden as Assessed by the Food Allergy Quality of Life-Parental Burden (FAQoL-PB):How Limited Would Your Ability to Participate in Social Activities That Involve Food be Because of Your Child's Food Allergy?
Description: as for outcome 11
Time Frame: Baseline and 4 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 20
score on a scale | 2.3 [1.2 to 3.4] | 1.7 [1.0 to 2.3]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT04512924/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT04512924/ICF_002.pdf